CLINICAL TRIAL: NCT03998683
Title: A Phase 3b, Multicenter, Interventional, Randomized, Placebo-controlled Study Investigating the Efficacy and Safety of Guselkumab for the Treatment of Palmoplantar-non-Pustular Psoriasis
Brief Title: A Study of Guselkumab for the Treatment of Palmoplantar-non-Pustular Psoriasis
Acronym: G-PLUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108611; 2018-003206-58 (EudraCT Number); CNTO1959PSO3013 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2019-06-25; First posted 2019-06-26 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guselkumab Group (Experimental): Participants will receive guselkumab 100 mg SC injections at Weeks 0, 4, 12 and placebo subcutaneous (SC) injection at Week 16 in double-blind phase followed by guselkumab 100 mg SC injections at Weeks 20, 28, 36, and 44 in open-label phase.
  Interventions: Drug: Guselkumab 100 mg; Drug: Placebo
- Placebo Group (Placebo Comparator): Participants will receive placebo SC injection at Weeks 0, 4, 12 and guselkumab 100 mg SC injection at Week 16 in double-blind phase followed by guselkumab 100 mg SC injection at Week 20, 28, 36, and 44 in open-label phase.
  Interventions: Drug: Guselkumab 100 mg; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab 100 mg — Guselkumab 100 mg will be administered as SC injection.
  Other Names: CNTO1959
Drug: Placebo — Placebo will be administered as SC injection.

SUMMARY:
The purpose of this study is to evaluate the efficacy of guselkumab for the treatment of palmoplantar psoriasis.

DETAILED DESCRIPTION:
Chronic plaque psoriasis is the most common form of psoriatic skin disease; however, there is growing evidence that other variants including scalp, nail, inverse, and palmoplantar psoriasis are prevalent, undertreated, and are correlated with an increased risk of psoriatic arthritis that may result in significant morbidity with functional impairment and greater impairment in quality of life. Therefore, the main aim of the study is to provide robust efficacy and safety data on guselkumab treatment for palmoplantar non-pustular psoriasis. The study comprises of a Screening Phase (4 Weeks [Week -4 to 0]), a Treatment Phase (up to Week 48) and a post-treatment follow-up phase (up to Week 56). Key efficacy assessments include physician assessments and patient-reported outcomes questionnaires. Safety evaluations will include 12-lead electrocardiogram at baseline, pregnancy testing and monitoring of vital signs at all visits and recording of adverse events throughout the study. Also, participants will be evaluated for signs and symptoms of active tuberculosis at all visits including follow-up visit. Biomarker assessments will include the evaluation of relevant markers in serum for all participants. The study will have an overall duration of 56 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Should have all the following: A confirmed diagnosis of moderate-to-severe palmoplantar-non-pustular psoriasis with palm and/or sole involvement and at least one plaque at a body site other than the palms and soles for at least 6 months, to confirm a diagnosis of chronic psoriasis; psoriatic area and severity index (PASI) score greater than or equal to (>=) 3 and less than (<) 10 at screening and at baseline; Palmoplantar Investigator Global Assessment (ppIGA) score >=3 at screening and at baseline
* Should be eligible to receive biological treatments; only participants who are naive to biological treatments can be included
* A woman of childbearing potential must have a negative urine pregnancy test at screening and at Week 0
* Agree not to receive a live virus or live bacterial vaccination during the study, or within 12 weeks after the last administration of study intervention
* Agree to avoid prolonged sun exposure and agree not to use tanning booths or other ultraviolet (UV) light sources from the first administration of study intervention through 12 weeks after the final dose of study intervention (Week 56)

Exclusion Criteria:

* Currently has palmoplantar pustulosis, pustular psoriasis, or any other forms other than plaque-type psoriasis (e.g, erythrodermic, guttate), or hyperkeratotic eczema
* Has current drug-induced psoriasis (eg, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* Has received prior systemic treatment with biological agents or Janus Kinase (JAK) inhibitors
* Has had prior exposure, known and reported intolerance to guselkumab or excipients, or ineligible to treatment with biological agents
* Is infected with human immunodeficiency virus (HIV, positive serology for HIV antibody)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Palmoplantar Pustulosis Psoriasis Area and Severity Index 75 (ppPASI75) Response at Week 16 | Week 16
  Percentage of participants who achieve ppPASI75 response, defined as improvement greater than or equal to (>=) 75 percent (%) in the ppPASI score at Week 16 will be reported. The ppPASI is an assessment tool based on the PASI that assesses erythema, pustules, desquamation and the extent of disease of the palms and/or soles.

SECONDARY OUTCOMES:
Change from Baseline in Body Surface Area (BSA) Score at Weeks 16, 24 and 48 | Baseline and Weeks 16, 24 and 48
  Change from baseline in BSA score at Week 16 will be reported in the guselkumab versus placebo group and at Weeks 24 and 48 will be reported separately for guselkumab and placebo-crossover groups by measuring the arithmetic mean of the affected skin surface.
Change from Baseline in absolute PASI Score at Weeks 16, 24 and 48 | Baseline, Weeks 16, 24 and 48
  Change from baseline in absolute PASI score at Week 16 will be reported in the guselkumab versus placebo group and at Weeks 24 and 48 will be reported separately for guselkumab and placebo-crossover groups.
Percentage of Participants Achieving PASI 75 Score at Weeks 16, 24 and 48 | Weeks 16, 24 and 48
  Percentage of participants achieving PASI 75 score (participants who achieve >=75% improvement in PASI score) at Weeks 16, 24 and 48 will be reported in guselkumab versus the placebo group. PASI is a common clinical tool used to measure the severity and extent of psoriasis. The PASI is an assessment tool based on the PASI that assesses erythema, pustules, desquamation and the extent of disease of the palms and/or soles.
Percentage of Participants Achieving PASI 90 Score at Weeks 16, 24 and 48 | Weeks 16, 24 and 48
  Percentage of participants achieving PASI 90 score (participants who achieve >=90 % improvement in PASI score) at Weeks 16, 24 and 48 will be reported in guselkumab versus the placebo group. PASI is a common clinical tool used to measure the severity and extent of psoriasis. The PASI is an assessment tool based on the PASI that assesses erythema, pustules, desquamation and the extent of disease of the palms and/or soles.
Percentage of Participants Achieving PASI 100 at Weeks 16, 24 and 48 | Weeks 16, 24 and 48
  Percenatge of participants who achieving PASI 100 score (participants who achieve >=100 % improvement in PASI score) at Weeks 16, 24 and 48 will be reported in guselkumab versus the placebo group. PASI is a common clinical tool used to measure the severity and extent of psoriasis. The PASI is an assessment tool based on the PASI that assesses erythema, pustules, desquamation and the extent of disease of the palms and/or soles.
Change from Baseline in Palmoplantar Quality-of-Life Instrument (ppQLI) Score at Weeks 16, 24 and 48 | Baseline and Weeks 16, 24 and 48
  Change from baseline in ppQLI score at Week 16 will be reported in the guselkumab versus placebo group and at Weeks 24 and 48 will be reported separately for guselkumab and placebo-crossover groups. ppQLI assesses relevant dimensions affected by palmoplantar psoriasis (pain/discomfort, functionality, and social/activity limitations) to assess quality of life.
Change from Baseline in Dermatology Life Quality Index (DLQI) Score at Weeks 16, 24 and 48 | Baseline and Weeks 16, 24 and 48
  Change from baseline in DLQI score at Week 16 will be reported in the guselkumab versus placebo group and at Weeks 24 and 48 will be reported separately for guselkumab and placebo-crossover groups. DLQI a 10-item questionnaire that can be used to assess overall quality-of-life.
Change from Baseline in European Quality of Life, 5-Dimension, 5-Level (EQ-5D-5L) Score at Weeks 16, 24 and 48 | Baseline and Weeks 16, 24 and 48
  Change from baseline in EQ-5D- 5L score at Week 16 will be reported in the guselkumab versus placebo group and at Weeks 24 and 48 will be reported separately for guselkumab and placebo-crossover groups. EQ-5D-5L is a standardized instrument to measure health-related quality of life.
Change from Baseline in Palmoplantar Investigator Global Assessment (ppIGA) Score at Weeks 16, 24 and 48 | Baseline and Weeks 16, 24 and 48
  Change from baseline in ppIGA score at Week 16 will be reported in the guselkumab versus placebo group and at Weeks 24 and 48 will be reported separately for guselkumab and placebo-crossover groups to assess psoriasis overall lesions.
Change from Baseline in Fingernail-Physician Global Assessment (f-PGA) Score at Weeks 16, 24 and 48 | Baseline and Weeks 16, 24 and 48
  Change from baseline in f-PGA score at Week 16 will be reported in the guselkumab versus placebo group and at Weeks 24 and 48 will be reported separately for guselkumab and placebo-crossover groups to assess fingernails separately for nail bed and nail matrix for signs of disease.
Percentage of Participants who Achieve ppPASI75 response at Weeks 24 and 48 | Weeks 24 and 48
  Percentage of participants who achieve ppPASI75 response, defined as improvement >=75% in the ppPASI score at Weeks 24 and 48 will be reported separately for guselkumab and placebo-crossover groups. The ppPASI is an assessment tool based on the PASI that assesses erythema, pustules, desquamation and the extent of disease of the palms and/or soles.
Percentage of Participants who Achieve ppPASI90 response at Weeks 24 and 48 | Weeks 24 and 48
  Percentage of participants who achieve ppPASI90 response (participants who achieve >=90 % improvement in the ppPASI score) at Weeks 24 and 48 will be reported separately for guselkumab and placebo-crossover groups. The ppPASI is an assessment tool based on the PASI that assesses erythema, pustules, desquamation and the extent of the affection of the palms and/or soles.
Percentage of Participants who Achieve ppPASI100 response at Weeks 24 and 48 | Weeks 24 and 48
  Percentage of participants who achieve ppPASI100 response (participants who achieve >=100 % improvement in the ppPASI score) at Weeks 24 and 48 will be reported separately for guselkumab and placebo-crossover groups. The ppPASI is an assessment tool based on the PASI that assesses erythema, pustules, desquamation and the extent of the affection of the palms and/or soles.
Change from Baseline in Work Productivity and Activity Impairment: Psoriasis (WPAI: PSO) Score at Weeks 16, 24 and 48 | Baseline and Weeks 16, 24 and 48
  Change from baseline in WPAI: PSO score at Week 16 will be reported in the guselkumab versus placebo group and at Weeks 24 and 48 will be reported separately for guselkumab and placebo-crossover groups. WPAI-PSO is a questionnaire which includes 6 questions to measure work productivity and activity impairment related to skin psoriasis.
Change from Baseline in Numerical Rating Scale: Pain (NRS:P) Score at Weeks 16, 24 and 48 | Baseline and Weeks 16, 24 and 48
  Change from baseline in NRS:P score at Week 16 will be reported in the guselkumab versus placebo group and at Weeks 24 and 48 will be reported separately for guselkumab and placebo-crossover groups. NRS:P is a self-administered scale that assess pain intensity in participants.
Number of Participants with Adverse Event (AEs) as a Measure of Safety and Tolerability | Up to 56 weeks
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (26):
- France (4):
  - CHU Bordeaux - Hopital St Andre, Bordeaux
  - Hôpital Edouard Herriot, Lyon
  - CHU de Nice Hopital de l Archet, Nice
  - Hopital Charles Nicolle, Rouen
- Germany (8):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - University Hospital Dresden, Dresden
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - MensingDerma research GmbH, Hamburg
  - Universitätsklinikum Schleswig Holstein Campus Lübeck, Lübeck
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitaetsklinikum Muenster, Münster
  - Centrovital, Witten
- Italy (4):
  - AOU di Cagliari, Cagliari
  - P.O. Vittorio Emanuele Azienda Ospedaliero Universitaria 'Policlinico Vittorio Emanuele', Catania
  - Ospedale Santa Chiara AO Universitaria Pisana, Pisa
  - Istituto Clinico Humanitas, Rozzano
- Spain (5):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. de Manises, Valencia
- United Kingdom (5):
  - Russell's Hall Hospital, Dudley
  - Chapel Allerton Hospital, Leeds
  - Barts Health NHS Trust, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency